CLINICAL TRIAL: NCT00044187
Title: The Assessment of a Anti-Obesity Agent for the Treatment of Olanzapine-Associated Weight Gain in Patients With Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder and Bipolar I Disorder
Brief Title: The Assessment of a Weight-Gain Agent for the Treatment of Olanzapine-Associated Anti-Obesity Agent in Patients With Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder, and Bipolar I Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5102; F1D-MC-HGJJ
Record Dates: First submitted 2002-08-21; First posted 2002-08-23 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Schizophrenia; Psychotic Disorders; Bipolar Disorder
Keywords: schizoaffective disorder; schizophreniform disorder; bipolar I disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — sibutramine

INTERVENTIONS:
Drug: Sibutramine

SUMMARY:
Olanzapine is currently marketed for the treatment of schizophrenia and acute manic episodes with bipolar 1 disorder. This Anti-obesity Agent is currently marketed for the management of obesity. In this study, the Anti-obesity Agent is being tested to see if it can treat weight gain that may be associated with taking olanzapine.

The purposes of this study are to determine the safety of olanzapine when given in combination with the Anti-obesity Agent and any side effects that might be associated with it and whether weight-gain agent can help treat weight gain that may be associated with taking olanzapine.

ELIGIBILITY:
Eligibility Criteria:

* You must be between the ages of 18 and 65. If you have reached your 66th birthday, you will not be able to participate.
* You must have been diagnosed with schizophrenia, schizoaffective disorder, schizophreniform disorder, or bipolar I disorder and be taking olanzapine.
* You must be able to visit the doctor's office as scheduled for the next 4 months.

Exclusion Criteria:

* You have a history of an illness that would cause weight loss or gain in the near future.
* You have taken remoxipride within the past 6 months.
* You are allergic to olanzapine or Anti-obesity Agent.
* You have uncontrolled high blood pressure, congestive heart failure, or have had a stroke.
* You have a serious medical illness, such as heart, liver, or kidney disease.
* You are pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2001-04; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - El Centro, California
  - Jacksonville, Florida
  - Miami, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Prairie Village, Kansas
  - Milford, Massachusetts
  - Clementon, New Jersey
  - Beachwood, Ohio
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Richmond, Virginia
  - Bellevue, Washington